CLINICAL TRIAL: NCT02243423
Title: Neonatal Acid-base Status After Elective Cesarean Delivery Under Spinal Anesthesia - a Comparison of Maternal Supine Horizontal Position Versus Left Lateral Table Tilt
Brief Title: Neonatal Acid-Base Status After C Section With Maternal Tilt vs. Supine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Richard M. Smiley, Virginia Apgar Professor of Anesthesiology at Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AAAO1851
Record Dates: First submitted 2014-09-06; First posted 2014-09-18 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Aortocaval Compression; Fetal Acidosis
Keywords: Aortocaval compression; Cesarean Section; Spinal Anesthesia; Phenylephrine
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SUPINE group (Experimental): The surgical table will remain horizontal after intrathecal (spinal) anesthesia injection for cesarean section. Choosing to position the patient supine is the intervention.
  Interventions: Procedure: SUPINE
- TILT group (Active Comparator): The surgical table will be turned to 15° of left lateral tilt after patients are laid supine after spinal anesthesia injection. The tilted group is the control group.
  Interventions: Procedure: TILT

INTERVENTIONS:
Procedure: SUPINE — Patients in the SUPINE group will receive spinal anesthesia for cesarean section in the sitting position, after which they will lay supine horizontal on the surgical table.
  A phenylephrine intravenous infusion will be titrated according to a set protocol, to maintain the systolic blood pressure at baseline.
  Arms: SUPINE group
Procedure: TILT — Patients will receive spinal anesthesia for cesarean section in the sitting position, after which they will lay on the surgical table, which will be tilted to the left by 15°.
  A phenylephrine intravenous infusion will be titrated according to a set protocol to maintain the systolic blood pressure at baseline.
  Arms: TILT group

SUMMARY:
This study aims to compare the neonatal acid-base status of women who remain supine horizontal, with women who are tilted to the left side by 15° during elective cesarean delivery at term under spinal anesthesia, with systolic BP maintained at baseline with a phenylephrine (PE) infusion. The null hypothesis is that the position of the patient (supine horizontal or tilted) during cesarean section will make no difference to neonatal wellbeing. The primary outcome will be the neonatal umbilical arterial base deficit (BD) at birth. The investigators will also examine the effects of maternal position during cesarean section under spinal anesthesia on maternal cardiac output (CO) and whether these changes have a correlation with the neonatal umbilical cord blood acid-base status. The secondary outcome will be the total phenylephrine dose requirement at 15 minutes after spinal injection.

DETAILED DESCRIPTION:
Methods: This will be a randomized trial structured as an equivalence trial. Subjects will be American Society of Anesthesiologists (ASA) I and II women aged ≥18 years, non-laboring, at term (>37 weeks gestation) with singleton pregnancies in cephalic presentation, scheduled for elective cesarean delivery under spinal anesthesia. Patients will receive spinal anesthesia for cesarean section in the sitting position, after which they will lay either supine horizontal or the surgical table will be tilted to the left by 15°, depending on the group to which they were randomized (SUPINE or TILT). An IV phenylephrine infusion will be administered to maintain systolic BP at baseline until delivery. A noninvasive hemodynamic monitoring system (NICOM, Cheetah Medical Inc., Vancouver, WA, USA) will continuously monitor CO and stroke volume. Neonatal umbilical vein and arterial blood gas results will be recorded.The null hypothesis is that the position of the patient (supine horizontal or tilted) during cesarean section will make no difference to neonatal wellbeing.

Statistical Design: The estimated sample size is the minimum number of study subjects required for rejecting the alternative hypothesis (i.e., accepting the null hypothesis). A significant difference between groups in the primary outcome, umbilical artery BD (which is a measure of fetal well being at the time of delivery and an indirect indicator of the adequacy of uteroplacental perfusion) would be of the order of magnitude of 2 mmol/L. Standard deviation of BD tends to be of this magnitude also. It would therefore require 22 subjects per group for 90% power to detect this magnitude of difference with alpha 0.05. Because BD is often not normally distributed, it is appropriate to increase sample size by 10-20%, and because the investigators have important secondary outcomes (PE usage, UA and UV pH, UV BD) the investigators intend to recruit 50 subjects per group to allow sufficient power for analysis of these secondary outcomes with appropriate correction for multiple comparisons, and allowing for 10% dropout. PE usage in the investigators previous study tends to have a standard deviation of about 30% of the mean, also roughly the magnitude of a clinically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II women aged ≥18 years
* Non-laboring
* At term (>37 weeks gestation) with singleton pregnancies in cephalic presentation
* Scheduled for elective cesarean delivery under spinal anesthesia.
* Maternal height will be between 150 - 180 cm and the body mass index (BMI)≤ 40 kg/m2.

Exclusion Criteria:

* Ruptured membranes
* Severe polyhydramnios or oligohydramnios
* Nonreassuring fetal heart rate
* Intrauterine growth restriction
* Abnormal lie - e.g. breech, transverse lie
* Multiple gestation
* Maternal comorbidities: hypertension, preeclampsia, other cardiovascular disease, renal failure, diabetes mellitus> 10 years, severe scoliosis or kyphosis, uterine abnormalities (e.g. large fibroids, bicornuate uterus)
* Medications - anti-hypertensive agents
* Current smoking or illicit drug use
* Failed spinal (sensory level < T6 after 15 minutes), need to convert to general anesthesia before delivery (exclusion from data analysis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Base deficit (umbilical artery) (mEq/L) | Within 2 hours of birth
  The primary outcome will be the neonatal umbilical arterial base deficit at birth.Neonatal umbilical vein and arterial blood gas results (these are routinely sent by the obstetric service at Columbia University Medical Center for all deliveries)

SECONDARY OUTCOMES:
Total phenylephrine dose (mg) | 15 minutes after spinal injection
  The secondary outcome will be the total phenylephrine dose requirement at 15 minutes after spinal injection. The phenylephrine (PE) infusion will be titrated to maintain the systolic arterial pressure (SBP) at baseline. If the SBP is at or above baseline, no PE will be administered. If SBP is 90-99% of baseline, PE infusion will be at 50 μg/min. If the SBP is 80-89% of baseline, PE will be 100 μg/min. If SBP is less than 80% of baseline, the infusion will be doubled to 200 μg/min. When SBP returns to more than 90% of baseline, the infusion will be returned to 50 μg/min. If the SBP remains < 80% of baseline after 1 minute at 200 μg/min, additional boluses of IV phenylephrine 80 μg may be given. If this regimen is unsuccessful at restoring SBP to >90% of baseline within 3 minutes, any other indicated maneuver may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Smiley, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian, Allen Hospital, New York, New York, United States

REFERENCES:
- [Background] Lee SW, Khaw KS, Ngan Kee WD, Leung TY, Critchley LA. Haemodynamic effects from aortocaval compression at different angles of lateral tilt in non-labouring term pregnant women. Br J Anaesth. 2012 Dec;109(6):950-6. doi: 10.1093/bja/aes349. Epub 2012 Oct 11. PMID 23059960
- [Background] Crawford JS, Burton M, Davies P. Time and lateral tilt at Caesarean section. Br J Anaesth. 1972 May;44(5):477-84. doi: 10.1093/bja/44.5.477. No abstract available. PMID 5044078
- [Background] Cluver C, Novikova N, Hofmeyr GJ, Hall DR. Maternal position during caesarean section for preventing maternal and neonatal complications. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD007623. doi: 10.1002/14651858.CD007623.pub3. PMID 23543552